CLINICAL TRIAL: NCT00848406
Title: An Observational Study to Obtain Normal Values of Inflammatory Variables in Induced Sputum, Exhaled Breath, and Bronchial Biopsies From Healthy Smoking and Non-smoking Individuals
Brief Title: A Study to Obtain Normal Values of Inflammatory Variables From Healthy Subjects
Acronym: NORM
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten van den Berge, Dr., University Medical Center Groningen
Other Study IDs: METc2009007
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Asthma; Copd
Keywords: bronchial; COPD; Asthma; sputum; biopsies
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, induced sputum, bronchial biopsies, brush and lining fluid, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: 30 individuals ≤ 40 years, who currently smoke ≥ 10 cigarettes/day and > 10 packyears
- 2: 30 individuals ≤ 40 years, who have not smoked during the last year, have never smoked for as long as a year (i.e. at least one cigarette per day or one cigar per week, AND have < 0.5 packyear.
- 3: 30 individuals above 40 years, who currently smoke ≥ 10 cigarettes per day, and > 20 packyears.
- 4: 30 individuals above 40 years, who have not smoked during the last year, have never smoked for as long as a year, and have < 0.5 packyear.

SUMMARY:
Smoking induces an inflammatory reaction in the airways which can ultimately result in persistent damage and the development of a Chronic Obstructive Pulmonary Disease (COPD). However, not all subjects who smoke end up with COPD. After long-term smoking, approximately 20% of subjects develop COPD. At this time, it is unclear why some subjects develop COPD, whereas others maintain a normal lung function.

In addition, smoking has important consequences in asthma. Patients with asthma who smoke have a more severe asthma and more often experience an asthma exacerbation. In addition, it has been shown that inhaled corticosteroids are less effective in smoking asthmatics.

With this research project, the researchers will investigate the effects of smoking on the airways. To this end, the researchers will compare markers of airway inflammation, lung function and symptoms between healthy smokers and non-smokers of varying age. In addition, the researchers will compare those healthy subjects with patients with asthma and COPD which are characterized in earlier studies.

ELIGIBILITY:
Inclusion Criteria:

* Have not smoked during the last year.
* Have never smoked for as long as a year.
* Have < 0.5 packyear.

Exclusion Criteria:

* Persons who used inhaled or oral corticosteroids during >5 years, or within the last 5 years.
* FEV1 <1.2 L
* A subject is not eligible to enter and participate if he does not agree that we inform his general practicioner about participation in the study and also about any unexpected finding during the study.
* Upper respiratory tract infection (e.g. colds), within 2 months.
* Pregnancy, or the possibility of being pregnant (i.e. women who do not use adequate anticonception as judged by the investigator).
* Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* Signs or symptoms of any other concomitant disease that, in the eyes of the investigator, can interfere with the study results.
* Known recent substance abuse (drug or alcohol).
* Claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-04; Primary Completion 2014-04 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
parameters for inflammation and remodelling in airway tissue | The duration of the study is estimated on 2 year

SECONDARY OUTCOMES:
Induced sputum, PC20 AMP, spirometrie, questionnaires, CT scan. | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berge, MD, PhD, Principal Investigator — University Medical C enter Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Nair GB, Galban CJ, Al-Katib S, Podolsky R, van den Berge M, Stevens C, Castillo E. An assessment of the correlation between robust CT-derived ventilation and pulmonary function test in a cohort with no respiratory symptoms. Br J Radiol. 2021 Feb 1;94(1118):20201218. doi: 10.1259/bjr.20201218. Epub 2020 Dec 15. PMID 33320729
- [Derived] Faiz A, Imkamp K, van der Wiel E, Boudewijn IM, Koppelman GH, Brandsma CA, Kerstjens HAM, Timens W, Vroegop S, Pasma HR, Boersma WG, Wielders P, van den Elshout F, Mansour K, Steiling K, Spira A, Lenburg ME, Heijink IH, Postma DS, van den Berge M. Identifying a nasal gene expression signature associated with hyperinflation and treatment response in severe COPD. Sci Rep. 2020 Oct 15;10(1):17415. doi: 10.1038/s41598-020-72551-0. PMID 33060632
- [Derived] Boudewijn IM, Faiz A, Steiling K, van der Wiel E, Telenga ED, Hoonhorst SJM, Ten Hacken NHT, Brandsma CA, Kerstjens HAM, Timens W, Heijink IH, Jonker MR, de Bruin HG, Sebastiaan Vroegop J, Pasma HR, Boersma WG, Wielders P, van den Elshout F, Mansour K, Spira A, Lenburg ME, Guryev V, Postma DS, van den Berge M. Nasal gene expression differentiates COPD from controls and overlaps bronchial gene expression. Respir Res. 2017 Dec 21;18(1):213. doi: 10.1186/s12931-017-0696-5. PMID 29268739
- [Derived] Telenga ED, Oudkerk M, van Ooijen PM, Vliegenthart R, Ten Hacken NH, Postma DS, van den Berge M. Airway wall thickness on HRCT scans decreases with age and increases with smoking. BMC Pulm Med. 2017 Feb 1;17(1):27. doi: 10.1186/s12890-017-0363-0. PMID 28143620
- [Derived] Hoonhorst SJ, Lo Tam Loi AT, Pouwels SD, Faiz A, Telenga ED, van den Berge M, Koenderman L, Lammers JW, Boezen HM, van Oosterhout AJ, Lodewijk ME, Timens W, Postma DS, Ten Hacken NH. Advanced glycation endproducts and their receptor in different body compartments in COPD. Respir Res. 2016 Apr 26;17:46. doi: 10.1186/s12931-016-0363-2. PMID 27117828
- [Derived] Hoonhorst SJ, Lo Tam Loi AT, Hartman JE, Telenga ED, van den Berge M, Koenderman L, Lammers JW, Boezen HM, Postma DS, Ten Hacken NH. Advanced glycation end products in the skin are enhanced in COPD. Metabolism. 2014 Sep;63(9):1149-56. doi: 10.1016/j.metabol.2014.06.006. Epub 2014 Jun 13. PMID 25034386
- [Derived] Hoonhorst SJ, ten Hacken NH, Lo Tam Loi AT, Koenderman L, Lammers JW, Telenga ED, Boezen HM, van den Berge M, Postma DS. Lower corticosteroid skin blanching response is associated with severe COPD. PLoS One. 2014 Mar 12;9(3):e91788. doi: 10.1371/journal.pone.0091788. eCollection 2014. PMID 24622644